CLINICAL TRIAL: NCT03564743
Title: Clinical Description of Spondylarthritis and Validation of Assessment of SpondyloArthritis International Society (ASAS) Criteria in West Indian Patients Seen in the Routine Consultation of Rheumatology.
Brief Title: Description of Spondylarthritis and Validation of ASAS Criteria in West Indian Patients Seen in Consultation of Rheumatology.
Acronym: SPACA
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 14/E/20
Record Dates: First submitted 2017-04-19; First posted 2018-06-21 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Spondyloarthritis
Keywords: Spondyloarthritis; ASAS criteria; Diagnosis criteria; Classification criteria
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Evaluation of ASAS criteria — Perform ASAS criteria at the time of physician diagnosis of chronic low back pain in rheumatological practice.

SUMMARY:
In 2004 an ASAS for the Assessment of SpondyloArthritis International Society decided to work to improve the criteria for classification of spondyloarthropathies to allow for early diagnosis, Nuclear magnetic resonance imaging (MRI). This approach led to the publication in 2009 of the classification criteria for spondylarthritis, in particular axial spondyloarthritis, as well as a proposal to modify the classification of criteria defined by Mr. Amor (AMOR) and European Spondylarthropathy Study Group (ESSG) criteria, taking into account the potential abnormalities visible in Magnetic Resonance Imaging Nuclear (MRI).

The performance (specificity, sensitivity, positive and negative predictive values) of the ASAS criteria was then prospectively tested on a sample of the Metropolitan Caucasian population and this systematic study allowed to estimate the performance of the ASAS criteria in the usual framework Of the French Liberal Rheumatology Consultation.

Note that this approach is exposed to a criticism of "circular" approach, indeed the expert who is the gold standard for the diagnosis, uses more or less consciously "criteria" based on the presence of such and such sign, then checks in this selected population the diagnostic validity of these signs.

However, no data on the performance of ASAS criteria are available in populations of African descent.

DETAILED DESCRIPTION:
Historically, spondyloarthritis is considered rare in these populations in the image of human Leukocyte Antigen B27 (HLA B27) which is observed only in 0.3% of individuals. Its presence determines the appearance of sacroiliitis - the cardinal sign of the disease - which is therefore rare. The recent contribution of MRI has changed investigators point of view and makes it possible to make the diagnosis in frequent situations but more atypical clinically.

In practice:

1. ASAS signs are not systematically found in the West Indies (sacroiliitis, uveitis, cervicitis, urethritis, inflammatory syndrome, HLAB27 ...)
2. Apart from cases associated with Chronic Inflammatory Bowel Disease (IBD), clinical panels are atypical and the ASAS criteria for little help
3. MRI imaging is used to correct diagnosis. It is therefore necessary to describe these patients and to study the interest of the ASAS criteria in this population On the other hand, the validation of the ASAS criteria is part of the recommendations of treatment of the SPA (spondyloarthritis) by the French Society of Rheumatology in 2014. Clearly a patient who does not validate these criteria does not have access to anti- tumor necrosis factor (TNF) biotherapies, effective but Expensive. Thus, it is not known whether West Indian patients validate these criteria or not, but it is clear that despite the large number of local SPAs, few receive anti-TNF biotherapies.

The investigators propose to describe a population of Caribbean spondyloarthritis through a cross-sectional observational study carried out with a sample of rheumatologist doctors in three sites (Martinique, Guadeloupe, French Guyana). The methodology of the cluster survey of physicians, with a systematic evaluation of the first patients seen in consultation (chronological selection) provides the best guarantee of representativeness.

The interest of this work is to reproduce exactly the methodology of a previous work carried out in a Caucasian population, validated and published, and thus be able to compare the value of the ASAS criteria between the Caucasian and Caribbean populations.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient seen in the usual framework of the consultation of rheumatology
* Patients consulting with:
* Presence or history of chronic low back pain (≥ 3 months) that started before the age of 45 with an onset of low back pain after 2005:
* Or with known sacroiliitis or asymmetric inflammatory rheumatism
* Or with chronic inflammatory bowel disease (Crohn, ulcerative colitis (RCH) ...) and associated inflammatory rheumatism
* Patients who received a lumbosacral MRI after 2005
* Patient not participating in a clinical trial

Exclusion criteria:

* Patient under 18 years of age
* Patient participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with presence or history of chronic low back pain (≥ 3 months) that started before the age of 45 with an onset of low back pain after 2005
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | September 2018
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks.
ASAS criteria | September 2018
  Assess the performance of ASAS criteria (sensitivity, specificity, positive predictive value, negative predictive value) at the time of physician's diagnosis of chronic low back pain in rheumatological practice (Evaluation of the concept of "diagnostic criteria" and Classification criteria).

SECONDARY OUTCOMES:
Assessment and comparison of ASAS performance against other classifications | September 2018
  Performance calculation of other classification systems (ESSG, Amor, New York modified): sensitivity, specificity, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: Michel MD De Bandt, Principal Investigator — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gran JT. An epidemiological survey of the signs and symptoms of ankylosing spondylitis. Clin Rheumatol. 1985 Jun;4(2):161-9. doi: 10.1007/BF02032287. PMID 3159533
- [Background] Dougados M, van der Linden S, Juhlin R, Huitfeldt B, Amor B, Calin A, Cats A, Dijkmans B, Olivieri I, Pasero G, et al. The European Spondylarthropathy Study Group preliminary criteria for the classification of spondylarthropathy. Arthritis Rheum. 1991 Oct;34(10):1218-27. doi: 10.1002/art.1780341003. PMID 1930310
- [Background] Amor B, Dougados M, Mijiyawa M. [Criteria of the classification of spondylarthropathies]. Rev Rhum Mal Osteoartic. 1990 Feb;57(2):85-9. French. PMID 2181618
- [Background] van der Linden S, Valkenburg HA, Cats A. Evaluation of diagnostic criteria for ankylosing spondylitis. A proposal for modification of the New York criteria. Arthritis Rheum. 1984 Apr;27(4):361-8. doi: 10.1002/art.1780270401. PMID 6231933
- [Background] Sieper J, van der Heijde D, Landewe R, Brandt J, Burgos-Vagas R, Collantes-Estevez E, Dijkmans B, Dougados M, Khan MA, Leirisalo-Repo M, van der Linden S, Maksymowych WP, Mielants H, Olivieri I, Rudwaleit M. New criteria for inflammatory back pain in patients with chronic back pain: a real patient exercise by experts from the Assessment of SpondyloArthritis international Society (ASAS). Ann Rheum Dis. 2009 Jun;68(6):784-8. doi: 10.1136/ard.2008.101501. Epub 2009 Jan 15. PMID 19147614
- [Background] Boy FN, Kayhan A, Karakas HM, Unlu-Ozkan F, Silte D, Aktas I. The role of multi-parametric MR imaging in the detection of early inflammatory sacroiliitis according to ASAS criteria. Eur J Radiol. 2014 Jun;83(6):989-996. doi: 10.1016/j.ejrad.2014.03.002. Epub 2014 Mar 22. PMID 24703519
- [Background] Arnett FC, Edworthy SM, Bloch DA, McShane DJ, Fries JF, Cooper NS, Healey LA, Kaplan SR, Liang MH, Luthra HS, et al. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis Rheum. 1988 Mar;31(3):315-24. doi: 10.1002/art.1780310302. PMID 3358796
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595